CLINICAL TRIAL: NCT02403284
Title: The Effect of Liraglutide on Dietary Lipid Induced Insulin Resistance in Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Phoenix VA Health Care System (U.S. Federal Agency)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 028; 1593855 (Other: Phoenix VA Health Care System IRBNet/VAIRRS)
Record Dates: First submitted 2014-11-03; First posted 2015-03-31 (Estimated); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Insulin Resistance
Keywords: insulin resistance; lipid metabolism; glucose metabolism; high fat diets
MeSH Terms: conditions — Insulin Resistance | interventions — Liraglutide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental): Liraglutide titration up to 1.8 mg/d over approximately 3 weeks
  Interventions: Drug: Liraglutide
- Sugar pill (Placebo Comparator): matching placebo and titration
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Liraglutide — Subcutaneous injection by patient
  Other Names: Victoza
  Arms: Liraglutide
Drug: Sugar Pill — Subcutaneous injection daily
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
In this research study, investigators will test the effects of an approved medication for diabetes,Liraglutide, to reduce insulin resistance that develops from eating a diet high in saturated fats.

DETAILED DESCRIPTION:
The specific aim of this study is to determine the ability of subacute liraglutide administration to protect against dietary lipid induced peripheral insulin resistance in non-diabetic subjects who have normal glucose tolerance. Recent data from our laboratory and others suggest that high fat meals, enriched with saturated fatty acids (SFA) in particular, have a unique and profound ability to induce rapid (in ≤ 24 hr) and profound onset of insulin resistance in humans. This is presumably mediated in part through delivery of lipids and lipid products generated during postprandial lipolysis into non-adipose tissue. This unique model therefore provides an excellent platform to test agents for their ability to inhibit dietary induced insulin resistance. As we and others have demonstrated the ability of GLP-1 receptor agonists to markedly suppress postprandial lipid elevations and to modify lipid metabolism, we hypothesize that liraglutide may be an effective agent to inhibit development of dietary induced insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years old
2. Body mass index (BMI) from 22 to 35 kg/m2
3. Normal glucose tolerance as determined by fasting blood glucose (< 100 mg/dl) and 75 gm glucose load (2 hr glucose <140 mg/dl)
4. Fasting triglyceride levels ≥ 75 mg/dl and <500 mg/dl

Exclusion Criteria:

1. Type 1 or 2 diabetes mellitus or a hemoglobin A1c value >6.5 mg/dl
2. Any diabetes medications in the past month, thiazolidinedione medications in the prior 3 months or prior regular use of insulin
3. Lactose intolerance or avoidance of dairy products
4. Creatinine > 2.0 mg/dl or other laboratory evidence of active disease, including hepatic enzyme elevation (AST or ALT) > 2.5 x normal and anemia (Hct < 35)
5. Known 'Nonalcoholic Fatty Liver Disease'
6. Malabsorption of fat or other nutrients, severe lactose intolerance or other significant gastrointestinal or pancreatic problems (including history of acute or chronic pancreatitis).
7. Recent history of nausea or vomiting
8. Acute bacterial or viral illness or evidence of other active infection in the past 4 weeks
9. Prior cardiovascular event, stable or unstable angina or other major illness in the past 6 months
10. Current regular use of anti-inflammatory medications or antioxidants in excess of a standard daily multi-vitamin, including over- the-counter medications and high dose salicylates (> 1 gm/ day)
11. Subjects receiving a lipid lowering medication must be on a stable dose for at least 6 weeks prior to participation.
12. Personal or family history of medullary thyroid carcinoma or in patients with multiple endocrine neoplasia 2
13. Ethanol consumption more than 4 oz day
14. Pregnancy, or lack of appropriate contraceptive use in premenopausal women (extremely rare in our older predominately male population)
15. Poorly controlled hypertension, systolic blood pressure (SBP) > 150 or diastolic blood pressure (DBP) > 90 on 2 or more occasions during screening visits. Subjects receiving blood pressure medication will be on a stable dosing for at least 6 weeks prior to participation.
16. BMI <22 and >35 kg/m2

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-03; Primary Completion 2021-04-28 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Whole Body Insulin Sensitivity (insulin suppression test) | 3 weeks
  An insulin suppression test will be measured before and approximately 3 weeks after each treatment phase. Key time frames for assessing steady state plasma glucose will be between 150 and 180 minutes during the insulin suppression test

SECONDARY OUTCOMES:
Postprandial lipid changes (area under the curve difference in triglyceride,total apolipoprotein B100, apolipoprotein B48, and apolipoprotein C3. | 3 weeks
  The major endpoints will be the area under the curve difference in triglyceride and free fatty acids between treatment arms on test day 1 and 2 following a standard meal. Other postprandial lipids will include total apolipoprotein B100, apolipoprotein B48, and apolipoprotein C3.
Postprandial changes in glucose metabolism (total and incremental area under the curve differences in glucose, insulin and glucagon) | 3 weeks
  total and incremental area under the curve differences in glucose, insulin and glucagon between treatment arms
Changes in adipose tissue insulin signaling pathway activation (compare insulin signaling pathway activity (e.g., Akt and insulin receptor phosphorylation) | 3 weeks
  Adipose tissue biopsy samples will be used to compare insulin signaling pathway activity (e.g., Akt and insulin receptor phosphorylation) in placebo and liraglutide treatment phases.
subcutaneous adipose tissue lipid intermediates (e.g., ceramide, diacylglycerol, acylcarnitine concentrations) | 3 weeks
  Adipose tissue biopsy samples will be used to compare lipid intermediates in placebo and liraglutide treatment phases.
skeletal muscle tissue lipid intermediates (e.g., ceramide, diacylglycerol, acylcarnitine concentrations) | 3 weeks
  skeletal muscle tissue samples will be used to compare lipid intermediates in placebo and liraglutide treatment phases.
Adipose tissue inflammation measures (e.g., interleukin (IL)-6, and -8, adiponectin, TNF-alpha, nuclear factor-kappa b, gene and protein expression) | 3 weeks
  Adipose tissue biopsy samples will be used to compare inflammation measures in placebo and liraglutide treatment phases.
Skeletal muscle inflammation measures (e.g., IL-6,8, TNF-alpha, nuclear factor-kappa b gene and protein expression) | 3 weeks
  skeletal muscle tissue samples will be used to compare inflammation measures in placebo and liraglutide treatment phases
Adipose tissue arteriole function (vasodilation measurement) | 3 weeks
  Adipose tissue biopsy samples will be used to isolate arterioles and measure ex vivo vascular function in placebo and liraglutide treatment phases.
Changes in skeletal muscle insulin signaling pathway | 3 weeks
  skeletal muscle biopsy samples will be used to compare insulin signaling pathway activity (e.g., Akt and insulin receptor phosphorylation) in placebo and liraglutide treatment phases.

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Reaven, MD, Principal Investigator — Carl T. Hayden Medical Research Foundation
Locations (1):
- Carl T. Hayden VA Medical Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Subject to VA regulation.